CLINICAL TRIAL: NCT01210950
Title: Autologous Transplantation of Bone Marrow Derived Mesenchymal Stem Cells in Distraction Osteogenesis in Patients With Limb-length Discrepancy
Brief Title: Distraction Osteogenesis in Limb-length Discrepancy With Mesenchymal Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Bone-006
Record Dates: First submitted 2010-09-25; First posted 2010-09-29 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2008-04

CONDITIONS: Leg Length Inequality
Keywords: distraction; osteogenesis; limb length discrepancy; callus
MeSH Terms: conditions — Leg Length Inequality; Callosities | interventions — Carboxylesterase; Reagins; Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cell and RPR recepients (Experimental): mesenchymal cells and plasma reach protein are injected to the callus center of short limb
  Interventions: Biological: cell and RPR injection

INTERVENTIONS:
Biological: cell and RPR injection — mesenchymal cells and Plasma reach Protein are injected to the callus center
  Other Names: cell therapy

SUMMARY:
Limb-length discrepancy can be due to many causes. These are divided into three groups: congenital (from birth), developmental (from a childhood disease or injury that slows or damages the growth plates), and posttraumatic (from a fracture that leads to shortening of the bone ends). There are three ways to equalize the limb-length discrepancy: use a shoe lift, shorten the long leg, lengthen the short leg. Most patients do not like wearing a lift greater than 2 cm (3/4 in). For discrepancies greater than 2 cm but less than 5 cm (2 in), shortening of the long leg can be considered, especially for tall persons. For growing children, this can be easily accomplished with a small, minimally invasive, uncomplicated procedure called epiphysiodesis.The investigators aim to evaluate if injection of bone marrow derived mesenchymal stem cells can shorten the treatment period by acceleration of bone regeneration during distraction osteogenesis.

DETAILED DESCRIPTION:
Distraction osteogenesis has been widely utilized to treat leg length discrepancy, deformity, nonunion, osteomyelitis, and bone loss. It has been found that most difficult conditions can be resolved with this method. In this study the aim is to observe if mesenchymal stem cell transplantation can enhance new bone formation during distraction osteogenesis.Patients undergo bone distraction , and about 2-3 weeks after distraction mesenchymal stem cell are injected at the callus site. In the case of large bone gap, mesenchymal stem cells are seeded on bone matrix and then placed in the bone gap. Each patient is assessed at interval time of 1 month for 6 months post surgery by X-Ray and at month 6 post surgery by computed tomography(CT) scans.

ELIGIBILITY:
Inclusion Criteria:

* both gender
* patient with limb-length discrepancy
* Age:18-65

Exclusion Criteria:

* Diagnosis of cancer,DM,CNS disorder,thyroid disease or respiratory disease
* Known allergic reaction to components of study treatment and/or study injection procedure
* Patients infected with hepatitis B,C or HIV
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
effect of mesenchymal cell transplantation to decrease limb inequal | 6 months
  evaluate the effect of mesenchymal cells transplantation with plasma reach protein in limb lengthening and decrease limb inequal

SECONDARY OUTCOMES:
improve life quality | 12 months
  mesenchymal cells transplantation improve patients life quality

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — President of Royan Institute; Mohammad reza Baghban Eslami Nejad, PhD, Study Director — Board scientific; Mohssen Emadeddin, MD, Principal Investigator — Orthopadic Investigator; Nasser Aghdami, MD,PhD, Principal Investigator — Head of Regenerative center
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Royan Institute — http://www.royaninstitute.org